CLINICAL TRIAL: NCT06165445
Title: Optimizing tDCS Protocol for Clinical Use in Patients With Major Depressive Disorder
Brief Title: Optimizing tDCS Protocol for Clinical Use in Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Leibniz Research Centre for Working Environment and Human Factors (Other); Neuroelectrics Corporation (Industry); Zanjan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, Technical University of Dortmund
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ifado-NE-ZUMS
Record Dates: First submitted 2023-11-24; First posted 2023-12-11 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Depressive Disorder; Cognitive Impairment; Psychiatric Disorder
Keywords: major depressive disorder; tDCS
MeSH Terms: conditions — Depressive Disorder; Cognitive Dysfunction; Mental Disorders; Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, parallel group trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: to secure investigator blinding, interventions were applied by independent investigators who were not involved in outcome measure ratings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional tDCS group (Active Comparator): The conventional tDCS group will receive 30 sessions of 20-minute stimulation at 2 mA intensities using standard electrodes (7 x 5 cm) over the target region
  Interventions: Device: transcranial direct current stimulation (tDCS)
- multi-channel tDCS group (Active Comparator): The multi-channel tDCS group will receive 30 sessions of 20-minute stimulation at 2 mA intensities using 7 electrodes (11 mm) over the target region
  Interventions: Device: multichannel transcranial direct current stimulation (tDCS)
- sham tDCS group (Placebo Comparator): The conventional tDCS group will receive 30 session of 20-minute placebo stimulation using standard electrodes (7 x 5 cm) over the target region
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — In tDCS, direct electrical currents at the intensity of interest (2 mA for example) are generated by an electrical stimulator and are noninvasively delivered to the scalp through a pair of saline-soaked sponge electrodes (7×5 cm) or via more than two but smaller round electrodes over the target regions.
  Arms: conventional tDCS group; sham tDCS group
Device: multichannel transcranial direct current stimulation (tDCS) — In multichannel tDCS, direct electrical currents at the intensity of interest (2 mA for example) are generated by an electrical stimulator and are noninvasively delivered to the scalp through more than two and smaller round electrodes over the target regions.
  Arms: multi-channel tDCS group

SUMMARY:
In this project, the efficacy of different tDCS protocols in major depression will be investigated. The tDCS protocols have already been investigated in humans, and results showed that stimulation intensity has a different effect on tDCS long-term aftereffects based on the human motor cortex model. The project has three major goals: first, we want to see if the differential outcome of tDCS dosage, as present in healthy populations, can be translated to patients with major depression. Second, we want to compare the efficacy of a multi-channel novel protocol with conventional tDCS modules. Lastly, we are interested in the safety and tolerability of optimized multi-channel. The project output will be an optimized tDCS protocol for major depression treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for a moderate-to-severe major depression, primarily by a DSM-5-based structured interview by a licensed psychiatrist, confirmed by score on Hamilton Rating Scale for Depression (HAMD)
* being 18-60 years old
* providing written informed consent
* If female, negative urine pregnancy test
* Treatment naïve or on a stable standard antidepressant regimen (including selective serotonin reuptake inhibitors (SSRIs), serotonin-noradrenaline reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MOAIs) or tricyclics (TCAs)) with no change in treatment 6-weeks prior to and during the tDCS intervention

Exclusion Criteria:

* smoker
* pregnancy
* alcohol or substance dependence
* history of seizure
* history of neurological disorder
* comorbid Schizophrenia Axis I disorder, bipolar disorder, substance abuse or dependence, dementia, personality disorder
* history of head injury
* currently receiving any form of Cognitive Behavioral Therapy, Dialectical Behavioral Therapy, or Acceptance and Commitment Therapy
* Presence of ferromagnetic objects in the body that are contraindicated for brain stimulation of the head (pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips, metallic prostheses, permanent eyeliner, implanted delivery pump, or shrapnel fragments)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
depressive symptoms | up to 3 months after the intervention
  the score on the the Montgomery-Åsberg Depression Rating Scale (MADRS)
depressive symptoms | up to 3 months after the intervention
  the score on the Hamilton Depression Rating Scale (HDRS). The HDRS is a multiple-item questionnaire designed for measuring adult depression and is administered by health care professionals. It is currently the most common depression measure used worldwide. Items on the HDRS are scored from 0 to 4 or 0 to 2 depending on the symptom assessed, with high scores indicating greater symptom pathology. scores typically ranging from 15 to 20 indicate a clinical level of depressive symptomatology
depressive symptoms | up to 3 months after the intervention
  the score on the Beck Depression Inventory (BDI-II). The BDI is a self-reported twenty-one questions about how the subject has been feeling in the last week, and each question has four answers ranging in intensity. Scoring 19 or higher on the BDI-II is considered moderate depression

SECONDARY OUTCOMES:
Working memory task | up to 1 month after the intervention
  Performance in the Spatial Working Memory (SWM) task, which is a recommended test for depression by Cambridge Cognition (CANTAB)
Attention task | up to 1 month after the intervention
  Performance in the Rapid Visual Information Processing (RVP) task, which is a recommended test for depression by Cambridge Cognition (CANTAB)
Emotion Recognition Task | up to 1 month after the intervention
  Performance in the Emotion Recognition Task (ERT), which is a recommended test for depression by Cambridge Cognition (CANTAB)
electroencephalogram (EEG) functional connectivity | up to 1 week after the intervention
  Change in the EEG functional connectivity in the frontal areas
electroencephalogram (EEG) power | up to 1 week after the intervention
  Change in the EEG alpha/theta/gamma power

CONTACTS AND LOCATIONS:
Locations (1):
- Zanjan University of Medical Sciences, Zanjan, Zanjan Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided